CLINICAL TRIAL: NCT01220284
Title: Dose-finding Study of Satraplatin in Combination With Oral Vinorelbine in Patients With Advanced Solid Tumors
Brief Title: Satraplatin and Vinorelbine in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Agennix (Industry); Pierre Fabre Laboratories (Industry)
Responsible Party: General Director, SENDO
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKSD00701; 2007DR2331 (Other: Swissmedic)
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; oral treatment; platinum compound; vinca alkaloid; drug combination
MeSH Terms: interventions — satraplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Satraplatin in combo with vinorelbine (Experimental): Escalating doses of satraplatin and oral vinorelbine in subsequent cohorts of 3-6 patients according to the type and severity grade of acute toxicities observed during cycle 1.
  The dose escalation process will be discontinued once the MTD is achieved.
  Interventions: Drug: Satraplatin in combo with vinorelbine

INTERVENTIONS:
Drug: Satraplatin in combo with vinorelbine — * Satraplatin (gelatin capsules) p.o. on days 1 to 5 (from 60 mg/m2 up to 80 mg/m2)
  * Vinorelbine (soft capsules) p.o. on days 1, 8 and 15 (from 60 mg/m2 up to 80 mg/m2) The treatment is repeated every 4 weeks.
  Other Names: - Satraplatin (codenamed JM216); - Vinorelbine, Navelbine

SUMMARY:
Vinorelbine (NVB) and platinum compounds are anticancer agents with broad spectrum of efficacy, clinically and preclinically proven synergism and only partially overlapping toxicities. Combinations with vinorelbine and platinum compounds with limited neurotoxicity are among the most used palliative regimens in a variety of solid tumors, including NSCLC, breast and cervical cancer. The oral platinum analogue satraplatin (SATRA) has been brought into clinical development because of the antitumor activity and toxicity comparable to those of carboplatin, together with a good acceptability of the oral administration.The recent availability of oral formulation of anticancer agents of proven efficacy in some indications is likely to become a valid option which could affect clinical daily management. The oral administration of vinorelbine and satraplatin might represent a reasonable option of palliative treatment in patients with advanced breast cancer, NSCL, GU or GY tumors for which a curative treatment can not be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/ cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative chemotherapy measures do not exist or are no longer effective.
2. Histological/cytological diagnosis of solid tumors in which treatment with oral vinorelbine and oral platinum compounds(preferentially breast, NSCL, GU or GY tumors) is medically indicated
3. Progressive disease (also in terms of tumor markers only, like CA 125 for ovary and PSA for prostate). No measurable disease is necessary.
4. Age 18-75 years
5. Prior chemotherapy of ≤ 2 lines for advanced disease
6. ECOG Performance Status < 2
7. Life expectancy of at least 3 months
8. The patient or his/her legal representative must be able to read, understand and provide written evidence of informed consent
9. Female patients must not be pregnant or lactating and must be willing to practice contraception. The effects of satraplatin on the developing human fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation.
10. Male patients that are not surgically sterile must be practicing a medically acceptable contraceptive regimen while on study treatment
11. Adequate organ function as defined by the following:

    * Serum creatinine < 1.5 mg/dl (< 132 umol/l)
    * ANC > 1500/microL
    * Hb > 10 g/dl
    * Platelet > 100,000/microL
    * Total bilirubin < ULN for the reference laboratory
    * AST and ALT and alkaline phosphatase (AP) must be within the designated range allowing for eligibility.

Exclusion Criteria:

1. Other chemotherapy treatment < 4 weeks prior to enrolment
2. Treatment with vinorelbine < 6 months from time of enrolment
3. Known resistance to platinum chemotherapy containing regimens (resistance is defined as PD while on treatment or a progression free interval < 6 months after completion of platinum therapy)
4. Known resistance to vinca alkaloids, treatment (including continuous infusion). Resistance is defined as PD while on treatment or a progression free interval < 6 months after completion of therapy
5. Hypersensitivity or allergic reactions to platinum compounds or vinorelbine
6. Radiotherapy involving > 30% of the active bone marrow
7. Radiotherapy < 4 weeks prior to enrolment
8. Pre-existing peripheral neuropathy > grade 1
9. Pre-existing CTCAE hearing loss or tinnitus ≥ grade 2
10. Metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, had a negative imaging study within 4 weeks of study entry, is clinically stable with respect to the tumor at the time of study entry, and is not receiving steroid therapy or taper
11. Patients who have not recovered (> grade 1) from the following toxicities of previous regimens before enrolment: fatigue, mucositis, nausea/vomiting, diarrhoea
12. Subject is currently enrolled in, or has not yet completed at least 30 days since ending other investigational device or drug trial(s) or is receiving other investigational agent(s)
13. Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, uncontrolled congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
14. Pre-existing malabsorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption
15. History of human immunodeficiency (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
16. Concurrent use of medications that inhibit cytochrome P450 3A4
17. History of bone marrow or major organ transplant
18. Prior high dose treatment with PBSC support

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) based upon study drug related dose limiting toxicities (DLTs) | 28 days
  The Maximum Tolerated Dose (MTD) is defined as the dose at which 2 out of 3 to 6 patients experience a DLT.

SECONDARY OUTCOMES:
Safety | whole study period
  Safety assessments include routine physical examinations and laboratory evaluations (blood cell counts, functional parameters and chemistry). Adverse events will be graded according to the NCI-CTCAE, Common Terminology Criteria for Adverse Events v.3.0.
Tumor response | every 2 months
  Tumor response in target and non-target lesions will be assessed according to the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Sessa, MD, Study Chair — Swiss Cancer Institute
Locations (2):
- Switzerland (2):
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Kantonspital Graubünden, Chur

REFERENCES:
- [Derived] Gallerani E, Cathomas R, Sessa C, Digena T, Bartosek AA, Dal Zotto L, von Moos R. A phase I study of the oral platinum agent satraplatin in combination with oral vinorelbine in patients with advanced solid malignancies. Onkologie. 2013;36(1-2):40-5. doi: 10.1159/000346671. Epub 2013 Jan 28. PMID 23429330